CLINICAL TRIAL: NCT00482911
Title: A Phase II Study of Combination Oral CC-5013 Lenalidomide (Revlimid™), Oral Sunitinib (Sutent™) and Low Dose Oral Metronomic Cyclophosphamide for the Treatment of Stage IV Ocular Melanoma
Brief Title: Lenalidomide, Sunitinib, and Cyclophosphamide in Treating Patients With Stage IV Eye Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator left the institute.
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Caryn Steakley, R.N., Deputy Clinical Director, Center for Cancer Research, National Institutes of Health Clinical Center (CC)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 070134; NCI-07-C-0134
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Results first posted 2012-11-14 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: Intraocular Melanoma; Malignant Conjunctival Neoplasm
Keywords: recurrent intraocular melanoma; metastatic intraocular melanoma; ciliary body and choroid melanoma, medium/large size; extraocular extension melanoma; iris melanoma; conjunctival melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — Cyclophosphamide; Lenalidomide; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1-lenalidomide & cyclophosphamide (Experimental): Participants first started on 2 Interventions (Dose A-QD) in Cycle 1, with 10 mg Lenalidomide (Len) once daily and 50 mg Cyclophosphamide (Cyc) once daily; 25 mg Sunitinib (Sun) was added once daily as a 3rd Intervention (Dose B-QD) from Cycle 2 onwards. Doses were adjusted in subsequent cycles depending on toxicity, including incremental step downs to 5/25/12.5 mg Len/Cyc/Sun once daily (Dose C-QD) or once every other day (Dose C-QOD).
  Interventions: Drug: cyclophosphamide; Drug: lenalidomide
- Cohort 2-sunitinib & cyclophosphamide (Experimental): 2 participants started Cycle 1 with Dose B as described above and had adjusted-dosing as described for Cohort 1. The remaining 7 participants began Cycle 1 with 10 mg Len, 25 mg Cyc and 12.5 mg Sun once daily (Dose D-QD). Doses were adjusted in subsequent cycles depending on toxicity, including step up to 10/50/12.5 mg Len/Cyc/Sun once daily (Dose E-QD) and step down to Dose D once every other day (Dose D-QOD).
  Interventions: Drug: cyclophosphamide; Drug: sunitinib malate

INTERVENTIONS:
Drug: cyclophosphamide — 25-50 mg by mouth once daily on days 1-28.
  Other Names: cytoxan
Drug: lenalidomide — 10 mg by mouth once daily on days 1-28.
  Other Names: revlimid
  Arms: Cohort 1-lenalidomide & cyclophosphamide
Drug: sunitinib malate — 12.5 - 25 mg by mouth once daily on days 1-28.
  Other Names: sutent
  Arms: Cohort 2-sunitinib & cyclophosphamide

SUMMARY:
RATIONALE: Lenalidomide may stop the growth of tumor cells by blocking blood flow to the tumor. Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving lenalidomide together with sunitinib and low doses of cyclophosphamide once a day may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving lenalidomide together with sunitinib and cyclophosphamide works in treating patients with stage IV eye melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with stage IV ocular melanoma treated with lenalidomide, sunitinib malate, and low-dose metronomic cyclophosphamide.

Secondary

* Determine the toxicity of this regimen in these patients.
* Determine the progression-free survival of patients treated with this regimen.
* Obtain blood, urine, and tissue samples from these patients, when easily accessible, to determine the effects of this regimen on pathways thought to have been modulated by this regimen in pre-clinical studies.

OUTLINE: This is nonrandomized, uncontrolled, open-label study.

Patients receive oral lenalidomide, oral sunitinib malate*, and oral low-dose cyclophosphamide once daily on days 1-28. Treatment repeats every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

NOTE: *Some patients will not receive sunitinib malate during course 1.

After completion of study treatment, patients are followed every 3 months for 2 years, every 4 months for 3 years and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ocular melanoma

  * Stage IV disease
* Measurable disease
* No active brain metastases

  * Patients with brain metastases must have had a complete excision or radiotherapy and remain asymptomatic with stable disease by magnetic resonance imaging (MRI) or computed tomography (CT) scan for ≥ 6 months

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy > 3 months
* Granulocyte count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance > 60 mL/min
* Bilirubin ≤ 2.0 mg/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 10 times upper limit of normal (ULN)
* Prothrombin time (PT)/partial thromboplastin time (PTT)/International Normalized Ratio (INR) normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use one highly effective method of contraception (with an additional method) or barrier methods of contraception for ≥ 4 weeks before, during, and for ≥ 4 weeks after completion of study therapy
* Ejection fraction normal by echocardiogram
* No acute, critical illness, including serious untreated infection
* No history of any of the following:

  * Unstable or newly diagnosed angina pectoris
  * Myocardial infarction within the past 6 months
  * New York Heart Association class II-IV heart disease
  * Congestive heart failure
  * Chronic obstructive lung disease requiring oxygen therapy
  * Chronic uncontrollable hypertension
  * Uncontrolled seizure activity
* No known human immunodeficiency virus (HIV) positivity
* No known hypersensitivity reaction to thalidomide, lenalidomide, sunitinib malate, or cyclophosphamide

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior therapy
* At least 4 weeks since prior surgery, chemotherapy (6 weeks for mitomycin C, nitrosoureas, or carboplatin), hormonal therapy, radiotherapy, or biological therapy
* No concurrent grapefruit or grapefruit juice
* No other concurrent antitumor therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-04 (Actual); Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven K. Libutti, MD, Principal Investigator — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Dosing Schedule 1: Len & Cyc
Arm/Group | Cohort 1-lenalidomide & Cyclophosphamide | Cohort 2-sunitinib & Cyclophosphamide
Started | 3 (All received Dose A-QD in cycle 1) | 0
Completed | 3 | 0
Not Completed | 0 | 0
Period: Dosing Schedule 1: Len, Cyc, & Sun
Arm/Group | Cohort 1-lenalidomide & Cyclophosphamide | Cohort 2-sunitinib & Cyclophosphamide
Started | 3 (All received Dose B-QD in cycle 2) | 2 (All received Dose B-QD in cycle 1)
Completed | 3 (1 stopped at Dose B-QD, 1 stopped at Dose C-QD, 1 stopped at Dose C-QOD) | 2 (1 stopped at Dose B-QD, 1 stopped at Dose C-QOD)
Not Completed | 0 | 0
Period: Dosing Schedule 2: Len, Cyc, & Sun
Arm/Group | Cohort 1-lenalidomide & Cyclophosphamide | Cohort 2-sunitinib & Cyclophosphamide
Started | 0 | 7 (All received Dose D-QD in cycle 1)
Completed | 0 | 7 (5 stopped at Dose D-QOD, 2 stopped at Dose D-QD (1 after first increasing to Dose E-QD))
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1-lenalidomide & Cyclophosphamide | Cohort 2-sunitinib & Cyclophosphamide | Total
Number analyzed (Participants) | 3 | 9 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 8 | 10
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (15.52) | 54.89 (6.44) | 57.27 (9.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 0 | 3 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 9 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 8 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 9 | 12

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Complete and Partial Response)
Description: Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response is the disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD.
Time Frame: 2 years
Population: Cohort 2 = 9 patients. Two patients received Dose B-QD in cycle 1 as outlined in participant flow. Seven patients received Dose D-QD in cycle 1 as outlined in participant flow.
Measure: Number; unit: Participants
Arm/Group | Cohort 1-lenalidomide & Cyclophosphamide | Cohort 2-sunitinib & Cyclophosphamide
Number analyzed (Participants) | 3 | 9
Participants
  Complete Response | 0 | 0
  Partial Response | 0 | 0

2. Primary Outcome: Toxicity
Description: Here is the number of participants with adverse events. For a detailed list of adverse events see the adverse event module.
Time Frame: 16 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Cohort 1-lenalidomide & Cyclophosphamide | Cohort 2-sunitinib & Cyclophosphamide
Number analyzed (Participants) | 3 | 9
Participants | 3 | 8

3. Primary Outcome: Overall Survival
Description: Time from date of on study to the date of death from any cause or last follow up
Time Frame: up to 16 months
Population: Overall survival is not the same as response, to obtain overall survival the investigator would have to follow patients until death, which the original investigator left the institution well before this outcome could be accomplished.
Arm/Group | Cohort 1-lenalidomide & Cyclophosphamide | Cohort 2-sunitinib & Cyclophosphamide
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Progression Free Survival
Description: Proportion of patients who progress or die after the start of treatment
Time Frame: up to 16 months
Population: as for outcome 3
Arm/Group | Cohort 1-lenalidomide & Cyclophosphamide | Cohort 2-sunitinib & Cyclophosphamide
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Changes in Gene Expression, Methylation and Protein Modification
Description: Ribonucleic acid (RNA), deoxyribonucleic acid (DNA) and protein obtained from blood, urine and/or tissue was to be evaluated for changes in gene expression, methylation and/or protein modification.
Time Frame: Baseline and end of treatment course 1 and 2, approximately 42 days
Population: as for outcome 3
Arm/Group | Cohort 1-lenalidomide & Cyclophosphamide | Cohort 2-sunitinib & Cyclophosphamide
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 16 months
Arm/Group | Cohort 1-lenalidomide & Cyclophosphamide | Cohort 2-sunitinib & Cyclophosphamide
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/9
Other Adverse Events (participants affected / at risk) | 3/3 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1-lenalidomide & Cyclophosphamide (N=3) | Cohort 2-sunitinib & Cyclophosphamide (N=9)
Infection (Infections and infestations) | 0 (0) | 1 (1) — (documented clinically or microbiologically) with grade 3 or 4 neutrophils (ANC < 1.0 x 10e9/L): lung pneumonia
Leukocytes (total WBC) (Investigations) | 0 (0) | 1 (1)
Neutrophils/granulocytes (ANC/AG) (Investigations) | 0 (0) | 1 (1)
Obstruction, GI: cecum (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1-lenalidomide & Cyclophosphamide (N=3) | Cohort 2-sunitinib & Cyclophosphamide (N=9)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (11)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 4 (7)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (3) | 2 (3)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Leukocytes (total WBC) (Investigations) | 3 (7) | 6 (11)
Lymphopenia (Investigations) | 1 (1) | 2 (2)
Mood alteration::Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mucositis/stomatitis (clinical exam)::Oral cavity (Gastrointestinal disorders) | 1 (1) | 1 (2)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Neutrophils/granulocytes (ANC/AG) (Investigations) | 3 (9) | 7 (16)
Pain: Abdomen NOS (Gastrointestinal disorders) | 1 (1) | 4 (5)
Pain::Head/headache (Nervous system disorders) | 1 (1) | 0 (0)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Pain::Neck (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Photosensitivity (Eye disorders) | 1 (1) | 0 (0)
Platelets (Investigations) | 1 (1) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (4) | 3 (4)
Rigors/chills (General disorders) | 2 (3) | 0 (0)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 2 (2) | 3 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 0 (0) | 2 (2)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Bilirubin (hyperbilirubinemia) (Investigations) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Edema: limb (General disorders) | 0 (0) | 1 (1)
Hemorrhage, GI::Rectum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Skin (cellulites)
Infection with normal ANC or Grade 1 or 2 neutrophils::Skin (cellulitis) (Infections and infestations) | 0 (0) | 1 (1)
Pain::Oral cavity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain::Oral gums (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No